CLINICAL TRIAL: NCT03529474
Title: Nonpharmacological Approach of Chronic Pain in Patients With Hemophilia: a Combined Approach From Psychology and Physiotherapy
Brief Title: Psychology and Physiotherapy Approach of Chronic Pain in Patients With Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/0320
Record Dates: First submitted 2018-03-14; First posted 2018-05-18 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Psychology; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychology and Physiotherapy group (Experimental): The psychological program consists of 4 sessions (2 hours each) comprising psychoeducation, training techniques of psychological management of pain and kinesiophobia resources The physiotherapy program consists of 3 domiciliary sessions per week, including physical exercise and stretching
  Interventions: Other: Psychology and Physiotherapy group
- Placebo Comparator: Control group (Placebo Comparator): Usual daily activities
  Interventions: Other: Placebo comparator: control group

INTERVENTIONS:
Other: Psychology and Physiotherapy group — Psychological program: 4 sessions,2 hours each,4 months
  * Psychoeducation.Influence of psychological factors on chronic pain: modulators of pain experience. Biopsychosocial model of pain.
  * Training techniques of psychological management of pain:Diaphragmatic Breathing and Progressive Muscle Relaxation to control vicious circle pain-tension-pain.
  * Kinesiophobia. Rational regulation of the activity level:Cognitive therapy (management of irrational believes about pain) and Organisation of time and reinforcement activities.
  Physiotherapy program:3 sessions per week,1 hour per session,4 months:
  * Aerobic exercise:walking, cycling
  * Warm-up: active ROM exercises of inferior and superior extremities (ISE)
  * Progressive resistance training with elastic bands of ISE
  * Stretching of ISE
  Arms: Psychology and Physiotherapy group
Other: Placebo comparator: control group — Control group Normal daily activities Usual daily activities
  Arms: Placebo Comparator: Control group

SUMMARY:
This study evaluates the clinical impact of a combined protocol with cognitive-behavioral intervention and physiotherapy adjuvant to the standard medical treatment in patients with haemophilia that suffer from chronic pain

DETAILED DESCRIPTION:
The purpose of this study is to improve the perception of the experience of chronic pain, as well as functionality and quality of life in hemophilic patients with chronic pain

Secondary objectives are:

* to change the perception that the patient has of their pain, to improve the coping strategies and to increase the perception of self-efficacy of patients in pain management.
* to increase the resources that allow a better self-regulatory of emotional, cognitive and competential of the pain experience, reverting in the emotional state of patients, particularly in levels of anxiety and depression.
* to improve functional capacity and musculoskeletal status.
* to improve quality of life.
* to determine whether changes / improvements are maintained over time 3 months after finishing the program

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of haemophilia A or B.
* Age between 18 and 60 years.
* Informed consent signed.
* Signs of arthropathy according to clinical criteria (score Gilbert) and / or radiological criteria (score Pettersson) in at least one of the six joints most commonly affected (ankles, knees or elbows)
* Chronic pain (CP) defined as persistent pain lasting at least six months and resistant to conventional medical therapy. It differs from the acute pain not only in its longer duration, but also sometimes persists even after the cause that produced it has disappeared.
* Absence of active coping strategies, understanding the concept of coping as those cognitive and behavioral efforts made by the individual in order to manage internal and external demands generated by their chronic pain condition and that involve a challenge to their potential individual resources.

Exclusion Criteria:

* Presence of inhibitor to FVIII or FIX.
* Another haemostatic defect.
* Patients with severe cognitive deficits with which it is not possible a cognitive psychological intervention.
* The inability to attend physiotherapy sessions for 12 consecutive weeks (7 supervised and 31 self-monitored)
* Surgical procedures performed 6 weeks prior or during the intervention protocol.
* Not acceptance or withdrawal of informed consent

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in Perceived Self-efficacy: Chronic Pain Self-Efficacy Scale Spainsh Version. (Martín-Aragon et al., 1999). | baseline, 4 months, 7 months
  The scale contain 3 Subscales: Self-efficacy in the control of symptoms (score 0-80); Self-efficacy in physical functioning (score 0-60) and Self-efficacy in pain management (score 0-50). Total Score: 0-190 and higher values represent a better outcome (more Self-Efficacy perceived).

SECONDARY OUTCOMES:
Quality of Life related with health | baseline, 4 months, 7 months
  Measured by a Specific questionnaire for Quality of Life related with health evaluation for adults with haemophilia (A36Haemophilia-QoL), which explores 9 areas. Subscales and score range: Physical health: 0-32; Daily activities: 0-16; Joints: 0-12; Pain: 0-8; Treatment satisfaction: 0-8; Difficulties treatment: 0-16; Emotional functioning: 0-20; Mental health: 0-12; Social activity: 0-20. Subscales are summed, with a total score from 0-144 and higher values represent a better outcome (more Quality of Life perceived).
Emotional status | baseline, 4 months, 7 months
  Patient's emotional state will be evaluated by Hospital Anxiety and Depression Scale (HAD), which assess the level of anxiety and depression. Subscales and score range are Anxiety (0-21) and Depression (0-21). Scoring: items of each subscale are summed, indicating: 0-7 normality, 8-10 probably case, 11-21 anxiety or depression clinical case. Higher values represent a worse outcome.
Nociceptive pain | baseline, 4 months, 7 months
  Nociceptive pain will be measured by the Visual Analog Scale for pain (VAS) from 0 to 10, where higher values represent a worse outcome.
Neuropathic pain | baseline, 4 months, 7 months
  Neuropathic pain evaluation by Pain Detect Questionnaire (Pain-Detect-Q-Spanish, with a total score 0-38, indicating: 0-12 absence of neuropathic pain; >12-18 doubtful diagnosis and >18-38 presence of neuropathic pain.
Kinesiophobia | baseline, 4 months, 7 months
  Kinesiophobia will be evaluated by Tampa Scale for Kinesiophobia (TSK-11SV) (Spanish adaptation. Gómez-Pérez, López-Martínez y Ruiz-Párraga, 2011). Scoring: Items are summed, with a total score from 11-44 and higher values represent a worse outcome (more pain interference in behavior).
Functional capacity: The Timed "Up & Go" test | baseline, 4 months, 7 months
  Timed "Up & Go" will be used to measure functional capacity. Less time to complete the test in seconds implies better outcome
Functional capacity: Sit-to-stand test | baseline, 4 months, 7 months
  Sit-to-stand test will be used to measure functional capacity. Less time to complete the test in seconds implies better outcome
Functional capacity: 2-minutes walk test | baseline, 4 months, 7 months
  Evaluation of functional capacity during walking by using 2 minutes walk test. More distance covered in 2 minutes implies better outcome.
Self-perceived functional capacity | baseline, 4 months, 7 months
  Impact of haemophilia on self-perceived functional abilities in adults measured by Haemophilia Activities List questionnaire (HAL). It contains 42 multiple choice questions in seven domains (Sum Score: 42-252). Normalized scores for the domains and the full questionnaire can also be obtained, being possible scores range from 0 to 100, where 0 represents the worst possible functional status and 100 the best possible functional status.
Active Range of Movement | baseline, 4 months, 7 months
  A digital goniometer will be used (Digital absolute Axis goniometer, Baseline evaluation instruments, White Plains, USA) for the measurement of active elbow, knee and ankle range of movement.
Joint health status | baseline, 4 months, 7 months
  Joint clinical evaluation of elbows, knees and ankles by using The Hemophilia Joint Health Score 2.1 (HJHS). The full score range goes from 0 to 124 points (0-20 points for each of the six joints evaluated, plus 4 points for the overall assessment of gait. 0 means no joint damage, whereas the higher the value, the higher the degree of arthropathy.

CONTACTS AND LOCATIONS:
Overall Officials: María García Dasí, Psych, Principal Investigator — Instituto de Investigación Sanitaria La Fe. Hospital Universitari i Politècnic La Fe
Locations (1):
- Instituto de Investigación Sanitaria La Fe. Hospital Universitari i Politècnic La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No